CLINICAL TRIAL: NCT06770322
Title: Comparison of Conventional and Manometry Measurement Methods in the Evaluation of Perioperative Laryngeal Edema by USG in Patients Undergoing Lumbar Stabilization Surgery
Brief Title: Comparison of the Effect of Two Methods on Laryngeal Edema in Endotracheal Cuff Inflation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fatih Sultan Mehmet Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Mustafa Berkehan Nizamlıoğlu, resident doctor, Fatih Sultan Mehmet Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: FSMTRH-MBN-01
Record Dates: First submitted 2024-12-28; First posted 2025-01-13 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-02

CONDITIONS: Spinal Stabilization
Keywords: ultrasonography; laryngeal edema; endotracheal cuff; lumbar spinal stabilization surgery
MeSH Terms: conditions — Laryngeal Edema | interventions — Congresses as Topic

STUDY DESIGN:
Intervention Model Description: two groups with a conventional and manometry group
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Conventional (Other): According to the clinician's own practice, the cuff of the endotracheal intubation tube will be manually inflated with the help of a syringe and the pressure will be measured with manometry and a note will be taken.
  Interventions: Procedure: Conventional
- Manometer (Experimental): The cuff pressure will be measured by manometry and the cuff of the endotracheal intubation tube will be inflated with 25-30 cmH2O.
  Interventions: Procedure: manometer

INTERVENTIONS:
Procedure: Conventional — According to the clinician's own practice, the cuff of the endotracheal intubation tube will be manually inflated with the help of a syringe and the pressure will be measured with manometry and a note will be taken.
  Arms: Conventional
Procedure: manometer — The cuff pressure will be measured by manometry and the cuff of the endotracheal intubation tube will be inflated with 25-30 cmH2O.
  Arms: Manometer

SUMMARY:
In this study, the investigators aimed to evaluate perioperative laryngeal edema in patients undergoing lumbar stabilization surgery in the pron position, which the investigators use in our routine anesthesia practice, by using conventional and manometry measurement methods and ultrasonography, which the investigators also use frequently in our routine, and to evaluate complications related to laryngeal edema in postoperative service follow-up.

DETAILED DESCRIPTION:
Prone position is the position in which the patient is laid on his/her abdomen, arms are turned to the sides and the head is turned to one side. Prone position is one of the most commonly used positions in different surgical procedures. Lumbar spinal surgeries (lumbar stabilization, lumbar disc herniation, etc.) are some of the types of surgical operations performed in the pron position. While giving pron position, the table and necessary materials are prepared. A thin pillow is placed under the head and the head is turned to one side. The arms are extended to the side or placed under the head. The abdomen is freed by placing a small support at the hip and shoulder level. Make sure that the eyes are closed to avoid eye pressure. In patients with large breasts and abdomen, a thin pillow is placed under the chest. The feet are supported with a pillow under the ankles. With this position under anesthesia, diaphragmatic movements are restricted as the body weight is placed on the abdominal wall, and the increase in intra-abdominal pressure makes venous return difficult. The breasts in women and genital organs in men may remain under pressure. Weight on bony structures and fingers may cause pressure trauma. These effects can be eliminated with a pillow placed at the shoulder and pelvis level and free movement of the abdomen is provided.

Hemodynamic and position-related complications can often be observed in patients operated in the pron position.

Complications related to the position itself include loss of vision, conjunctival redness ischemic orbital compartment syndrome, nerve damage, abdominal compartment syndrome, acute glaucoma, diplopia, pneumocephalus, shoulder dislocation, endotracheal tube obstruction, facial edema, enteral nutrition intolerance, accidental extubation and small bowel obstruction may be observed. Hemodynamic complications include decreased venous return due to increased intra-abdominal pressure and consequently decreased stroke volume, increased sympathetic response, increased heart rate, increased systemic and pulmonary vascular resistance and decreased left ventricular compliance due to increased intrathoracic pressure. Laryngeal edema may be observed due to compression on the face, jaw and neck and also due to compression of the intubation tube cuff on the tracheal wall and may constitute a risk factor for the development of postextubation stridor after extubation. Laryngeal edema may cause sore throat, cough, dysphonia, dysphagia and even reintubation due to narrowed airway in the patient after extubation, which is seen in the definition of postextubation stridor.

One of the drawbacks of this position in patients to be given general anesthesia is the decrease in airway safety. There is a possibility of tube dislodgement, displacement and kinking during and after the patients are turned to pron position. Therefore, patients should be intubated with a spiral tube, the tube location should be verified and fixed, and the tube location should be verified again after turning to the pron position.

The ideal pressure of the cuff of the intubation tube is 25-30 cmH2O when measured with a cuff manometer. The conventional method, which has been the practice for years, i.e. inflating the intubation cuff with a syringe according to the clinician's own practice, may cause edema in the tracheal wall and larynx and even tracheal necrosis after a while if the cuff is inflated too much. It has been demonstrated that if the pressure of the intubation tube cuff exceeds 30 cm H2O, the blood flow in the tracheal mucosa starts to decrease and if it exceeds 50 cm H2O, ischemic damage develops.

Tracheal damage and laryngeal edema may develop due to high cuff pressure. To prevent this, attention should be paid to measurement of cuff pressure by manometry. The recent development of ultrasonography, which is one of the imaging methods, has facilitated the prevention of laryngeal edema and edema-related complications in patients.

The cuff lowering test is a simple method used to predict the occurrence of stridor due to laryngeal edema after extubation. The test is performed by lowering the cuff and measuring the expired tidal volume after a few breaths. The leak is calculated as the difference between the tidal volume with and without the cuff deflated. However, since the cuff remains deflated throughout the respiratory cycle, a volume of gas may also leak during inspiration and therefore this method measures the total leakage consisting of the inspiratory and expiratory component. While airway stenosis was measured with the cuff lowering test before ultrasonography was introduced into practice, with the introduction of ultrasonography into clinical practice, the possibility of laryngeal edema and complications in patients has become predictable and measures have been taken accordingly. With ultrasonography, laryngeal edema development can be observed in patients by measuring the air column width after intubation and before extubation in the transverse axis with a linear probe over the patient's cricothyroid membrane.

Evaluation of laryngeal edema in patients operated in the pronated position with the cuff lowering test and the effect of cuff inflation with the cuff lowering test, conventional method and manometry on laryngeal edema have been shown in studies. However, in literature search, the participants did not find any comparison of the effect of cuff inflation with ultrasonography on laryngeal edema in patients who were operated in the pron position and in patients who were operated in the pron position. In routine anesthesia practice, the participants use the pron position and ultrasonography, which belongs to clinic, in accordance with the preferences of the individuals. In this study, the participants aimed to evaluate perioperative laryngeal edema in patients undergoing lumbar stabilization surgery in the pron position, which the participants use in our routine anesthesia practice, by using conventional and manometry measurement methods and ultrasonography, which we also use frequently in our routine, and to evaluate complications related to laryngeal edema in postoperative service follow-up. This study will be conducted with a total of 60 patients between the ages of 18-65 who will undergo lumbar stabilization surgery by neurosurgery between December 2024 and June 2025 under elective conditions in Fatih Sultan Mehmet Training and Research Hospital after obtaining ethics committee approval. Patients will be divided into 2 groups. One group will be the Conventional group (C) and the other group will be the Measurement with Manometry (M) group.

Patients with a history of direct laryngoscopy and biopsy, microlaryngoscopic surgery, tonsillectomy, adenoidectomy, surgery in the oral cavity such as soft palate, oropharynx, hypopharynx, larynx and trachea; allergy, asthma, reflux, upper respiratory viral or fungal infections and cancer surgery; receiving radiotherapy to the neck region; and patients who had more than one intubation attempt in the previous year, patients who will undergo emergency surgery, patients with advanced cardiac, renal, pulmonary and hepatic insufficiency, and patients who did not give consent to participate in the study will be excluded from the study.

Patients admitted to the operating room will receive standard monitoring including electrocardiogram (ECG), peripheral oxygen saturation (SpO2) monitoring, invasive arterial monitoring, intake and output fluid monitoring, perioperative vasopressor use and Sedline for monitoring brain functions for monitoring the depth of anesthesia.

Following monitoring, anesthesia induction will be provided with 2-2.5 mg/kg iv propofol, 2 mcg/kg iv fentanyl and 0.6 mg/kg iv rocuronium after premedication with midazolam. After adequate muscle relaxation, patients will be intubated by direct laryngoscopy using an orotracheal spiral tube of appropriate size. In intubation, the cuff of the endotracheal intubation tube of the conventional (K) group will be manually inflated according to the clinician's own practice and the inflated value will be measured by manometry and noted. In the manometry measurement group, the cuff of the endotracheal intubation tube will be inflated with 25-30 cmH2O. After intubation, the patient's air column width will be measured in the transverse axis using the linear probe of ultrasound, which the participants routinely use in clinic, from the cricothyroid membrane area of the patient. Patients will be transferred to the anesthesia device and mechanical ventilation will be applied with end-tidal carbon dioxide values between 35-40 mmHg, volume control mode, tidal volume 8 ml/kg, peep: 5, respiratory rate 10-14 /min. Patients will be carefully turned to the pron position and the head of the patients will be placed on the pron position pillow in such a way that there is no eye, nose and throat pressure. For maintenance of anesthesia, desflurane at a concentration of 4-6% in 40% O2-Air and 0.05-0.2 mcg/kg/min iv remifentanil infusion will be administered to all patients with a fresh gas flow of 2 lt/min. Anesthetic drugs will be titrated so that heart rate (HR) and/or mean arterial pressure (MAP) will not change more than 20% of the baseline value and Sedline PSI value will be between 25-50. For postoperative analgesia, 1 g paracetamol and 1 mg/kg tramadol and for postoperative nausea prophylaxis, 4 mg ondansetron will be administered iv. When skin sutures are applied, desflurane will be turned off, fresh gas flow will be increased to 8 l/min in both groups and 80% O2-air will be continued. The patient will be turned from pron position to supine position at the end of the operation. After the patients are turned to supine position, air column width will be measured and recorded before extubation. Patients with spontaneous respiratory effort will be given 2 mg/kg sugammadex iv to reverse neuromuscular blockade. Patients with adequate respiratory effort will be extubated and taken to the recovery unit when consciousness is clear, muscle strength is restored and hemodynamically stable. During the operation, routine hemodynamic parameters such as SpO2, invasive arterial pressure, heart rate, respiratory rate, respiratory rate, end-tidal CO2, inspiratory-expiratory oxygen and anesthetic gas concentrations, airway pressures (Ppik, Pplato), invasive arterial pressure and Sedline PSI values will be monitored and recorded at the same time with the measurement times. In addition, the presence of nausea, vomiting and tremor will be recorded at recovery. Patients with Aldrete score ≥ 8 will be transferred to the ward.

Air column width measurements will be performed by anesthesiologists using the ultrasound device of our own clinic and will be performed after intubation before turning to pron position and before extubation after turning from pron position to supine position and the ratio of pre-extubation value to post-intubation value will be recorded. Air column measurements will be performed after lowering the endotracheal cuff after aspirating the oral secretions of the patients. After the measurements are made, the cuff of the endotracheal tube will be inflated with the help of manometry at the same pressure.

Patients will be questioned about postoperative cough, dyspnea, dysphagia, dysphonia, dysphonia, sore throat and facial edema due to postoperative laryngeal edema at the 4th, 8th and 24th postoperative hours.

ELIGIBILITY:
Inclusion Criteria:

* Patients who will undergo lumbar spinal surgery under general anesthesia under elective conditions
* Patients aged 18-65 years, included in the ASA I-III group
* Patients whose consent has been obtained

Exclusion Criteria:

* Patients under 18 years of age, over 65 years of age, included in the ASA IV-V group
* Patients with a history of surgery in the oral cavity, including direct laryngoscopy and biopsy, microlaryngoscopic surgery, tonsillectomy, adenoidectomy, soft palate, oropharynx, hypopharynx, larynx and trachea,
* Patients with a history of allergies, asthma, reflux, upper respiratory viral or fungal infections and cancer surgeries,
* Patients receiving radiotherapy to the neck who had multiple intubation attempts in the previous year,
* Patients undergoing emergency surgery,
* Patients with advanced cardiac, renal, pulmonary and hepatic failure,
* Patients who did not give consent to participate in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-07-10 (Actual)

PRIMARY OUTCOMES:
Measurement of airway column width | through study completion, an average of 6 months
  Measurement of the effect of conventional and manometry methods on air column width by ultrasonography. With ultrasonography, laryngeal edema development can be observed in patients by measuring the air column width after intubation and before extubation in the transverse axis with a linear probe over the patient's cricothyroid membrane

SECONDARY OUTCOMES:
Detection of complications due to postoperative laryngeal edema | It will be evaluated at PACU 5th minute and postoperative 4, 8, 24th hours
  Detection of cough, dyspnea, dysphagia, dysphonia, dysphonia, facial edema that may occur after surgery for laryngeal edema.

CONTACTS AND LOCATIONS:
Overall Officials: Arzu Yildirim Ar, As Prof, Study Director — Fatih Sultan Mehmet Training and Research Hospital
Locations (1):
- Fatih Sultan Mehmet Training and Research Hospital, Istanbul, Atasehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kwee MM, Ho YH, Rozen WM. The prone position during surgery and its complications: a systematic review and evidence-based guidelines. Int Surg. 2015 Feb;100(2):292-303. doi: 10.9738/INTSURG-D-13-00256.1. PMID 25692433
- [Background] Oliveira VM, Weschenfelder ME, Deponti G, Condessa R, Loss SH, Bairros PM, Hochegger T, Daroncho R, Rubin B, Chiste M, Batista DC, Bassegio DM, Nauer Wda S, Piekala DM, Minossi SD, Santos VF, Victorino J, Vieira SR. Good practices for prone positioning at the bedside: Construction of a care protocol. Rev Assoc Med Bras (1992). 2016 May-Jun;62(3):287-93. doi: 10.1590/1806-9282.62.03.287. PMID 27310555
- [Background] Shriver MF, Zeer V, Alentado VJ, Mroz TE, Benzel EC, Steinmetz MP. Lumbar spine surgery positioning complications: a systematic review. Neurosurg Focus. 2015 Oct;39(4):E16. doi: 10.3171/2015.7.FOCUS15268. PMID 26424340
- [Background] Bentsianov BL, Parhiscar A, Azer M, Har-El G. The role of fiberoptic nasopharyngoscopy in the management of the acute airway in angioneurotic edema. Laryngoscope. 2000 Dec;110(12):2016-9. doi: 10.1097/00005537-200012000-00007. PMID 11129012
- [Background] Manohar N, Ramesh VJ, Radhakrishnan M, Chakraborti D. Haemodynamic changes during prone positioning in anaesthetised chronic cervical myelopathy patients. Indian J Anaesth. 2019 Mar;63(3):212-217. doi: 10.4103/ija.IJA_810_18. PMID 30988536
- [Background] AK AK, Cascella M. Post-Intubation Laryngeal Edema. 2023 Jul 4. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK560809/ PMID 32809644
- [Background] Seegobin RD, van Hasselt GL. Endotracheal cuff pressure and tracheal mucosal blood flow: endoscopic study of effects of four large volume cuffs. Br Med J (Clin Res Ed). 1984 Mar 31;288(6422):965-8. doi: 10.1136/bmj.288.6422.965. PMID 6423162
- [Background] Prinianakis G, Alexopoulou C, Mamidakis E, Kondili E, Georgopoulos D. Determinants of the cuff-leak test: a physiological study. Crit Care. 2005 Feb;9(1):R24-31. doi: 10.1186/cc3012. Epub 2004 Nov 29. PMID 15693963
- [Background] El-Baradey GF, El-Shmaa NS, Elsharawy F. Ultrasound-guided laryngeal air column width difference and the cuff leak volume in predicting the effectiveness of steroid therapy on postextubation stridor in adult. Are they useful? J Crit Care. 2016 Dec;36:272-276. doi: 10.1016/j.jcrc.2016.07.007. Epub 2016 Jul 16. PMID 27468680
- [Background] Abdel Wahab Abdelsattar Saleh Mohammad, Yara Ayman Iskandarani, Wael Mohammed Mossa, Maher A sheriff, Mohamrd Hamdi Alqassas. Comparative Study between Cuff Leak Test and Laryngeal U/S for Detection of Post Extubation Oedema in Prone Position Patient with General Anesthesia. J. Med. Chem. Sci., 2023, 6(11) 2686-2698.